CLINICAL TRIAL: NCT06630975
Title: Resident at AlAzhar University Assuit
Brief Title: Hemiepiphysiodesis by Eight Plate Versus Osteotomy in the Management of Pediatric Coronal Knee Deformities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Osama Hamdy, Mohamed Osama Hamdy, Al-Azhar University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEPVOMPCKD
Record Dates: First submitted 2024-09-20; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Genu Varum
MeSH Terms: conditions — Genu Varum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Comparative Study between Growth guided Correction By ( 8 Plate ) (Experimental): Coronal angular deformities of lower limb in children are a common finding in pediatric orthopedic surgery.
  Interventions: Device: Hemiepiphysiodesis; Procedure: Eight-Plates first described by Stevens are simple to use; Device: Hemiepiphysiodesis by eight Plate
- Clinical ,Radiological of Comparison the Result of Growth guided Correction to Osteoclasis in mana (Other): These angular deformities can be idiopathic in origin, or they can emerge secondary to congenital and acquired abnormalities. Valgus deformities in excess of 10* can cause anterior knee pain, circumduction gait, and occasionally patellofemoral instability. Varus deformities may result in lateral thrust, ligamentous laxity, and a waddling gait , meniscal tears, collateral ligament laxity, cartilage degeneration, and early osteoarthritis due to gradual mechanical axis disruption
  Interventions: Device: Hemiepiphysiodesis; Procedure: Eight-Plates first described by Stevens are simple to use; Device: Hemiepiphysiodesis by eight Plate
- Comparison the Result of Growth guided Correction to Osteoclasis (Active Comparator): These angular deformities can be idiopathic in origin, or they can emerge secondary to congenital and acquired abnormalities. Valgus deformities in excess of 10* can cause anterior knee pain, circumduction gait, and occasionally patellofemoral instability. Varus deformities may result in lateral thrust, ligamentous laxity, and a waddling gait , meniscal tears, collateral ligament laxity, cartilage degeneration, and early osteoarthritis due to gradual mechanical axis disruption
  Interventions: Device: Hemiepiphysiodesis; Procedure: Eight-Plates first described by Stevens are simple to use; Device: Hemiepiphysiodesis by eight Plate
- Genu Varum (Active Comparator): These angular deformities can be idiopathic in origin, or they can emerge secondary to congenital and acquired abnormalities. Valgus deformities in excess of 10* can cause anterior knee pain, circumduction gait, and occasionally patellofemoral instability. Varus deformities may result in lateral thrust, ligamentous laxity, and a waddling gait , meniscal tears, collateral ligament laxity, cartilage degeneration, and early osteoarthritis due to gradual mechanical axis disruption
  Interventions: Device: Hemiepiphysiodesis; Procedure: Eight-Plates first described by Stevens are simple to use; Device: Hemiepiphysiodesis by eight Plate

INTERVENTIONS:
Device: Hemiepiphysiodesis — 8 plate
Procedure: Eight-Plates first described by Stevens are simple to use — fewer complications in terms of implant loosening and fracture can be expected.Good results as well as low rebound and complication rates have been recorded
Device: Hemiepiphysiodesis by eight Plate — Extraperiosteal eight plate insertion

SUMMARY:
Coronal angular deformities of lower limb in children are a common finding in pediatric orthopedic surgery.These angular deformities can be idiopathic in origin, or they can emerge secondary to congenital and acquired abnormalities. Persistent coronal plane deformities around knee (genu varum/valgum) could lead to meniscal tears, collateral ligament laxity, cartilage degeneration, and early osteoarthritis due to gradual mechanical axis disruption

DETAILED DESCRIPTION:
Eight-Plates first described by Stevens are simple to use .Moreover, owing to the flexible screw/plate connection, fewer complications in terms of implant loosening and fracture can be expected.Good results aswell as low reboundand complication rates have been recorded for the first series of cases

ELIGIBILITY:
Inclusion Criteria:

* Growth plate still open at Time of Surgery

Exclusion Criteria:

* Epiphyseal plate involved in trauma resulting in a bridging callus formation,

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Comparative Study Between Growth Guided Correction By ( 8 Plate ) and Corrective Osteoclasis in Management of Coronal Deformity of Lower Limb in Children | 1 year
  Coronal angular deformities of lower limb in children are a common finding in pediatric orthopedic surgery.These angular deformities can be idiopathic in origin, or they can emerge secondary to congenital and acquired abnormalities. Persistent coronal plane deformities around knee (genu varum/valgum) could lead to meniscal tears, collateral ligament laxity, cartilage degeneration, and early osteoarthritis due to gradual mechanical axis disruption

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammad Osama Hamdy, Asyut, Egypt